CLINICAL TRIAL: NCT01389531
Title: Evaluation of the Efficacy and Safety of the HCPA-1 Silicone Stent in the Treatment of Central Airway Obstructions
Brief Title: Efficacy and Safety Evaluation of HCPA-1 Silicone Stent in the Treatment of Central Airway Obstructions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ORTESE 10-0515; ORTESE HCPA-1 (Other Grant/Funding Number: Ministerio da Saude/MS)
Record Dates: First submitted 2011-06-17; First posted 2011-07-08 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Tracheobronchomalacia
MeSH Terms: conditions — Tracheobronchomalacia | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stents (Other): All recruited patients will be receiving a stent during a rigid bronchoscopy procedure.
  Interventions: Procedure: Rigid bronchoscopy

INTERVENTIONS:
Procedure: Rigid bronchoscopy — The HCPA-1 silicone stent available in the following dimensions (diameter x length in mm): 9x30, 9x50, 11x30, 11x50, 13x30, 13x50, 14x30, 14x50, 16x50, 16x70, 18x50 and 18x70 will be inserted through rigid bronchoscopy in patients who presented the criteria to participate in the study.
  Other Names: stents

SUMMARY:
The aim of the study is, primarily, evaluate the safety of the use of the silicone stent HCPA-1 in patients with clinically significant tracheal and/or bronchial stenosis. Secondarily, this study aims to evaluate the efficacy of the use of the silicone stent HCPA-1 who are in the same conditions described above and also estimate the costs the use of these silicone stents involve.

DETAILED DESCRIPTION:
* It is a prospective multicenter clinical study, not controlled, with evaluation of clinical variables before and after the intervention (insertion of one or more silicone stents in the trachea or bronchi and main or intermediate bronchus by rigid bronchoscopy under general anesthesia).
* 110 patients, both genders, will be followed for one year, total of 8 visits, in order to evaluate the safety of the procedure of stent insertion.

It is allowed to include patients for whom it is indicated the combination of treatments (eg, electrocoagulation followed by stent placement) - full anticoagulation or severe disturbance of coagulation. (Includes: use of any anticoagulant, by oral, intravenous or subcutaneous administration with full intention of coagulation / therapy; coagulopathy with INR> 2.0 or aPTT [KTTP]> 1.5 times control or platelet count <50000). Note: The use of antiplatelet drugs (aspirin, clopidogrel, ticlopidine) is allowed.

- The HCPA-1 silicone stent is made of biocompatible silicone, medical grade, via injection process in the matrix using different densities of the same material for a set of prostheses with rigid and flexible variables; available in the following dimensions (diameter x length in mm): 9x30, 9x50, 11x30, 11x50, 13x30, 13x50, 14x30, 14x50, 16x50, 16x70, 18x50 and 18x70. Requires specific surgical (applicator) for insertion.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate in the study by signing (the patient or family member/ legal guardian) of the Informed Consent Form;
* 18 years old or more;
* clinically significant stenosis (symptomatic or about to become symptomatic) for the trachea, main bronchus or intermediate bronchus, which can be treated with the stent implement.

Exclusion Criteria:

* clinical or absolute anesthesic contraindication of the rigid bronchoscopy under general anesthesia;
* constitutional or acquired anatomic limitations that prevent the rigid bronchoscopy;
* another indication of exclusive preferential treatment modality for stenosis (surgery, radiotherapy, chemotherapy, other). Note: It is allowed to include patients for whom it is indicated the combination of treatments (eg, electrocoagulation followed by stent placement);
* full anticoagulation or severe disturbance of coagulation. (Includes: use of any anticoagulant, by oral, intravenous or subcutaneous administration with full intention of coagulation / therapy; coagulopathy with INR> 2.0 or aPTT [KTTP]> 1.5 times control or platelet count <50000). Note: The use of antiplatelet drugs (aspirin, clopidogrel, ticlopidine) is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2011-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measurement of Safety | 1 year
  three main adverse events will be followed:
  * migration of the stent;
  * granuloma formation;
  * accumulation of secretion

SECONDARY OUTCOMES:
Improvement in Dyspnea using a Dyspnea score as a measurement of Efficacy | 1 year
  MMRC dyspnea score will be used to measure the improvement of the patient's respiratory condition

CONTACTS AND LOCATIONS:
Overall Officials: Amarilio V Macedo, Postdoc, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (9):
- Brazil (9):
  - Hospital Universitario Getulio Vargas, Manaus, Amazonas
  - Hospital Universitario de Brasilia, Brasília, Federal District
  - Hospital das Clínicas de Goiania, Goiânia, Goiás
  - Hospital Universitario Antonio Pedro, Niterói, Rio de Janeiro
  - Hospital do Cancer I, Rio de Janeiro, Rio de Janeiro
  - Centro de Ciencias da Saude, Natal, Rio Grande do Norte
  - HCPA Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Paulo, São Paulo, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo

REFERENCES:
- [Background] Saueressig MG, Sanches PR, Macedo Neto AV, Moreschi AH, Oliveira HG, Xavier RG. Novel silicone stent to treat tracheobronchial lesions: results of 35 patients. Asian Cardiovasc Thorac Ann. 2010 Dec;18(6):521-8. doi: 10.1177/0218492310388428. PMID 21149399